CLINICAL TRIAL: NCT05083871
Title: Cognitive Appraisals and Team Performance Under Stress in Simulated Trauma Care
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Manchester Metropolitan University (Other); Humanitas Clinical and Research Center (Other); Azienda Sanitaria Universitaria Friuli Centrale (Other)
Responsible Party: Sponsor
Other Study IDs: 798-2021-OSS-AUSLBO
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Trauma; Stress, Emotional; Cognitive Change
Keywords: Medical simulation, Cognitive appraisal, Stress psychology
MeSH Terms: conditions — Wounds and Injuries; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Learners of the European Trauma Course: Learners attending the European Trauma Course
  Interventions: Other: European Trauma Course

INTERVENTIONS:
Other: European Trauma Course — Structured learning program specifically focused on Trauma management. The course provides frontal lessons, workshops for the technical skills and simulated scenarios.
  Please see https://www.erc.edu/courses/european-trauma-course for additional details

SUMMARY:
Medical teams work in demanding situations that are often uncertain, changeable and require accurate decision-making, skilled movement and coordinated action. How teams perform matters for patient outcomes. In addition to medical expertise, how individuals and the team collectively respond and manage the psychological stress of the situation has a significant impact on performance. One approach, which attempts to explain the facilitating and debilitating effects of stress on performance is the biopsychosocial model of challenge and threat. A challenge state occurs when perceived personal resources meet or exceed the situation's demands, whereas threat occurs when demands exceed resources. Challenge states have been consistently associated with improved performance in a range of environments and activities, including medical settings. In a recent study conducted during a national simulation-based training event for residents (the SIMCUP Italia 2018) it was found that a high level of resources is associated with better performance until demands become very high. The present study builds on previous work to explore how challenge and threat states are linked to performance. It includes a more recently developed and robust measure of demands and resource appraisals. In addition, secondary aims include the exploration of how psychological variables, specifically cognitive anxiety, somatic anxiety, self-confidence and social identity (connection with other members of the medical team) are linked to challenge and threat and performance. Understanding the psychological determinants of performance in critical care can provide the basis for individual and team-based interventions to improve critical care team performance.

ELIGIBILITY:
Inclusion Criteria:

* Learners of the European Trauma Course in Italy

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include all the learners attending the European Trauma Course in Italy, independently from their previous work experience and educational background
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Performance in simulated emergency trauma care | 3 days
  Composite outcome measure taking into account both technical and non technical skills evaluation from the course instructors

SECONDARY OUTCOMES:
participants' perceptions of task demands vs. personal resources | 3 days
  Evaluation of the evolution of the participants' perceptions of task demands vs. personal resources throughout the course
mental readiness | 3 days
  Evaluation of the evolution of the participants' mental readiness throughout the course
Social identity | 3 days
  Evaluation of the evolution of the participants' social identity throughout the course

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Unità Sanitaria Locale, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendes WB, Major B, McCoy S, Blascovich J. How attributional ambiguity shapes physiological and emotional responses to social rejection and acceptance. J Pers Soc Psychol. 2008 Feb;94(2):278-91. doi: 10.1037/0022-3514.94.2.278. PMID 18211177
- [Background] Tomaka J, Blascovich J, Kibler J, Ernst JM. Cognitive and physiological antecedents of threat and challenge appraisal. J Pers Soc Psychol. 1997 Jul;73(1):63-72. doi: 10.1037//0022-3514.73.1.63. PMID 9216079
- [Background] Blascovich J, Mendes WB, Hunter SB, Salomon K. Social "facilitation" as challenge and threat. J Pers Soc Psychol. 1999 Jul;77(1):68-77. doi: 10.1037//0022-3514.77.1.68. PMID 10434409
- [Background] Turner MJ, Jones MV, Sheffield D, Slater MJ, Barker JB, Bell JJ. Who thrives under pressure? Predicting the performance of elite academy cricketers using the cardiovascular indicators of challenge and threat states. J Sport Exerc Psychol. 2013 Aug;35(4):387-97. doi: 10.1123/jsep.35.4.387. PMID 23966448
- [Background] Vine SJ, Freeman P, Moore LJ, Chandra-Ramanan R, Wilson MR. Evaluating stress as a challenge is associated with superior attentional control and motor skill performance: testing the predictions of the biopsychosocial model of challenge and threat. J Exp Psychol Appl. 2013 Sep;19(3):185-94. doi: 10.1037/a0034106. PMID 24059821
- [Background] Carenzo L, Braithwaite EC, Carfagna F, Franc J, Ingrassia PL, Turner MJ, Slater MJ, Jones MV. Cognitive appraisals and team performance under stress: A simulation study. Med Educ. 2020 Mar;54(3):254-263. doi: 10.1111/medu.14050. Epub 2020 Feb 7. PMID 32034800
- [Background] Mendes WB, Gray HM, Mendoza-Denton R, Major B, Epel ES. Why egalitarianism might be good for your health: physiological thriving during stressful intergroup encounters. Psychol Sci. 2007 Nov;18(11):991-8. doi: 10.1111/j.1467-9280.2007.02014.x. PMID 17958714
- [Background] Franc JM, Verde M, Gallardo AR, Carenzo L, Ingrassia PL. An Italian version of the Ottawa Crisis Resource Management Global Rating Scale: a reliable and valid tool for assessment of simulation performance. Intern Emerg Med. 2017 Aug;12(5):651-656. doi: 10.1007/s11739-016-1486-7. Epub 2016 Jun 16. PMID 27312510
- See also: European Trauma Course official site — https://www.erc.edu/courses/european-trauma-course